CLINICAL TRIAL: NCT07156812
Title: Custom-Made 3D PEEK Plates Versus 3D Titanium Plates in Mandibular Angle Fracture Fixation: A Randomized Controlled Clinical Trial
Brief Title: Custom-Made 3D PEEK for Fixation of Mandibular Angle Fractures.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00010556-12/2021
Record Dates: First submitted 2025-08-28; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Mandibular Angle Fracture; Three Dimensional; Polyetheretherketone
Keywords: mandibular angle fracture; PEEK; three-dimensional plate fixation

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Investigator
Masking Description: Patients were allocated in a 1:1 ratio using an on-site computer software system with concealed allocation through sequentially numbered, opaque, sealed envelopes (SNOSE). Group A was treated with custom made 3D PEEK plates and Group B with 3D titanium plates.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with recent mandibular angle fractures managed with custome made 3D PEEK plate (Experimental): custome made 3D PEEK plate
  Interventions: Device: Custome made 3D PEEK plate
- patients with recent mandibular angle fractures managed with 3D Titanium plates (Experimental): 3D Titanium plates
  Interventions: Device: 3D Titanium plate

INTERVENTIONS:
Device: Custome made 3D PEEK plate — Custome made 3D PEEK plate
  Arms: patients with recent mandibular angle fractures managed with custome made 3D PEEK plate
Device: 3D Titanium plate — Pre-bent 3D Titanium plate
  Arms: patients with recent mandibular angle fractures managed with 3D Titanium plates

SUMMARY:
This investigation aimed to determine the clinical and radiographic efficacy of patient-specific, custom-made 3D PEEK plates in comparison with 3D titanium plates for the management of mandibular angle fractures.

DETAILED DESCRIPTION:
Eighteen patients with recent mandibular angle fractures indicated for open reduction and internal fixation were randomly allocated into two groups. The study group (n = 9) underwent fixation with custom-made 3D PEEK plates, while the control group (n = 9) received prebent 3D titanium plates adapted on virtually reduced models. Follow-up extended to 12 weeks. Clinical parameters included operative time, postoperative occlusion, interfragmentary stability, wound healing, and bite force recovery. Radiographic evaluation was conducted using computed tomography scans acquired immediately postoperatively and at 12 weeks, assessing fracture healing and mean bone density.

ELIGIBILITY:
Inclusion Criteria:

* patients with recent mandibular angle fracture adults without gender predilection who agreed to follow-up, fractures requiring open reduction and internal fixation, medically fit for general anesthesia

Exclusion Criteria:

* medically compromised patients, fractures with infection, pathological or old fractures, completely edentulous patients, comminuted fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Radiographic evaluation for the assessment of mean bone density at the fracture line [Time Frame: 12 weeks] | 12 weeks
  Mean bone density at the fracture line was assessed using Computed Tomography (CT) scan in Hounsfield Units (HU)
Bite force recovery. | 12 weeks
  bite force recovery measured by a Piezoresistive force transduce sensor: FlexiForce A201 sensor (FlexiForce sensor, by Tekscan Boston, MA, USA. www.tekscan.com)

SECONDARY OUTCOMES:
Clinical evaluation for interfragmentary stability. | 12 weeks
  Intra-fragmentary mobility was evaluated by bimanual palpation at the fracture site
clinical evaluation of wound healing | 14 days
  Wound healing is graded according to Southampton wound-grading system
Clinical evaluation of postoperative occlusion | 12 week
  By checking the maximal intercuspal position (centric occlusion) to ensure proper occlusal relationship including molar relation, canine relation and midline centralization

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all data will be de-identified to protect the participant data. patients signed an informed consent for the use of their medical records and data for study
Supporting Information: SAP

REFERENCES:
- [Derived] Kamal AO, Shaaban AM, Shokry MM, Abdelhamed IM. Custom-made 3D PEEK plates versus 3D titanium plates for mandibular angle fracture fixation: a randomized clinical trial. BMC Oral Health. 2026 Jan 30. doi: 10.1186/s12903-025-07646-z. Online ahead of print. PMID 41618317